CLINICAL TRIAL: NCT06542939
Title: Scaling Telehealth Models to Improve Co-morbid Diabetes and Hypertension in Immigrant Populations (Phase II)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01192-2; 5R01MD018528-02 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus Type II; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Workers (CHW) treatment group (Experimental): There is a 6-month intervention period immediately following recruitment. Participants enrolled in the intervention will complete 5 educational sessions and attend 2 one-on-one virtual meetings.
  Interventions: Behavioral: Integrated CHW Intervention
- Control group (Active Comparator): The control participants will complete only the first educational session. The control arm will receive usual care from their primary care physician (PCP) during the first 12 months of data collection. After 12 months they will be invited to attend remaining group sessions.
  Interventions: Behavioral: CHW Session 1 Only

INTERVENTIONS:
Behavioral: Integrated CHW Intervention — Participants will undergo all 5 group-based health education sessions on hypertension and diabetes management and provide culturally and linguistically tailored health information and resources. There will be two one-on-one virtual meetings, up to 9 follow-up phone calls to engage in goal-setting activities regarding changes to health behaviors, medication adherence, or other issues related to diabetes prevention as identified jointly by patient and CHW. Participants will develop with the CHW and receive a copy of their long-term and short-term Participant Action Plan. Referrals to other services available in the community (i.e. exercise classes, social services, mental health, tobacco cessation, etc.
  Arms: Community Health Workers (CHW) treatment group
Behavioral: CHW Session 1 Only — Participants will attend only the first group-based health education session on hypertension and diabetes management.
  Arms: Control group

SUMMARY:
The purpose of this study is to test the effectiveness and implementation process of a culturally and contextually tailored telehealth-based community health workers (CHW) led coaching intervention for hypertension control among South Asian patients with co-morbid Diabetes Mellitus type II (DMII) and hypertension. The primary aims are to test the effectiveness of a CHW-led telehealth intervention compared to usual care, and using Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) and Consolidated Framework for Implementation Research (CFIR), examine the reach, adoption, fidelity, and maintenance of the intervention within clinical and community settings.

ELIGIBILITY:
Inclusion Criteria:

* identified as of South Asian ethnicity
* at least 21 years of age
* a diagnosis of diabetes
* a diagnosis of hypertension
* an uncontrolled BP reading (>130/80mmHg) in the last 6 months

Exclusion Criteria:

* under the age of 21
* Women who are pregnant
* Type 1 diabetes or diabetes secondary to other conditions (e.g. steroid-induced, pancreatic insufficiency, or chemotherapy-induced)
* inability to perform unsupervised physical activity

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants achieving BP control, defined as <130/80 mmHg | Month 6
  The primary outcome will be the proportion of eligible patients at a practice site to achieve BP control (130/80 mmHg) at six months.

SECONDARY OUTCOMES:
Percent of participants achieving BP control, defined as <130/80 mmHg | Month 12
  The primary outcome will be the proportion of eligible patients at a practice site to achieve BP control (130/80 mmHg) at twelve months.
Change from Baseline in hemoglobin A1c (HbA1c) levels at Month 6 | Baseline, Month 6
  Change in HbA1c will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in HbA1c levels at Month 12 | Baseline, Month 12
  Change in HbA1c will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in Body mass index (BMI) at Month 6 | Baseline, Month 6
  Change in BMI will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in BMI at Month 12 | Baseline, Month 12
  Change in BMI will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in Systolic blood pressure (SBP) at Month 6 | Baseline, Month 6
  Change in SBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in SBP at Month 12 | Baseline, Month 12
  Change in SBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in Diastolic blood pressure (DBP) at Month 6 | Baseline, Month 6
  Change in DBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Change from Baseline in DBP at Month 12 | Baseline, Month 12
  Change in DBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: laura.wyatt@nyulangone.org . The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to laura.wyatt@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.